CLINICAL TRIAL: NCT00952575
Title: A Phase II, Open-label, Randomised, Dose-finding Study to Compare the Efficacy (in Terms of Clearance of RhD-positive RBCs) and Safety of LFB-R593, a Monoclonal Anti-RhD Antibody vs a Polyclonal Anti-RhD Immunoglobulin in Healthy RhD Negative Volunteers
Brief Title: Dose-finding Study of LFB-R593, A Monoclonal Anti-RhD Antibody, in Healthy RhD Negative Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: ADNC-0726
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Healthy
Keywords: Prevention of foeto-maternal allo-immunisation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- polyclonal anti-D immunoglobulin (Active Comparator)
  Interventions: Drug: polyclonal anti-D immunoglobulin
- Monoclonal anti-D immunoglobulin (Experimental)
  Interventions: Drug: monoclonal anti-D immunoglobulin

INTERVENTIONS:
Drug: polyclonal anti-D immunoglobulin — single injection of 300 µg
  Arms: polyclonal anti-D immunoglobulin
Drug: monoclonal anti-D immunoglobulin — Comparison of different dosages of LFB-R593
  Arms: Monoclonal anti-D immunoglobulin

SUMMARY:
This phase II study is designed to demonstrate the ability of LFB-R593 to effectively eliminate exogenously-administered RhD-positive red blood cells from the circulation of an RhD-negative individual, thereby preventing RhD-alloimmunisation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy RhD-negative volunteers
* Males and definitively sterile females
* No prior sensitization to RhD antigen

Exclusion Criteria:

* Healthy RhD-positive volunteers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Clearance of RhD-positive red blood cells | within 2 weeks after RBC injection

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kornicke, Principal Investigator — Parexel
Locations (1):
- Parexel Early Phase Clinical Unit, Berlin, Germany